CLINICAL TRIAL: NCT03629691
Title: A Retrospective Study for Patients With Lung Metastatic Advanced Gastric Cancer or NSCLC Treated With Apatinib
Brief Title: Study for Patients With Lung Metastatic Advanced Gastric Cancer and NSCLC Treated With Apatinib
Status: Completed | Type: Observational
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Other Study IDs: OG317
Record Dates: First submitted 2018-07-04; First posted 2018-08-14 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: Gastric Cancer Metastatic to Lung; Lung Cancer
Keywords: Cavitation; PFS
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- gastric cancer lung metastatic: One of the study tumors.Between February 1, 2015 and May 19, 2018, 356adult patients with gastric adenocarcinoma, multiline chemotherapy failure and lack of standard treatment, received oral apatinib 250 mg daily at the Affiliated Hospital of Qingdao University, of them, 110 patients with lung metastasis. 28 patients with lung cavitation
  Interventions: Other: lung cavitation
- NSCLC: One of the study tumors.Between February 1, 2015 and May 19, 2018, 77 adult patients with primary lung cancer, multiline chemotherapy failure and lack of standard treatment, received oral apatinib 250 mg daily at the Affiliated Hospital of Qingdao University. 30 of 77 were squamous cell carcinoma and 47 of 77 were adenocarcinoma. 28 patients with lung cavitation.
  Interventions: Other: lung cavitation

INTERVENTIONS:
Other: lung cavitation — apatinib treated patients developed lung cavitation

SUMMARY:
The primary end point was progression-free survival (PFS), secondary end points included duration of locoregional control (LRC), overall survival (OS), quality of life and safety. For metastatic lung cancer, LRC is the local control of metastatic lung tumor here.

DETAILED DESCRIPTION:
Between February 1, 2015 and May 19, 2018, 433 adult patients with gastric adenocarcinoma, lung adenocarcinoma and lung squamous cell carcinoma, multiline chemotherapy failure and lack of standard treatment, received oral apatinib 250 mg daily at the Affiliated Hospital of Qingdao University. Histologically proven were identified retrospectively using the Clinical Research Information Systems (CRIS) database. All patients were with Karnofsky performance status ≥70% or an Eastern Cooperative Oncology Group performance status of 0 to 1, with stable hepatic, hematologic, and renal functions. Cardiac disease and hemorrhagic disease were excluded. All patients had pre-therapy chest computed tomography (CT) prior to apatinib treatment, and follow-up chest CT at least every 4 weeks. The primary end point was progression-free survival (PFS), secondary end points included duration of locoregional control (LRC), overall survival (OS), quality of life and safety. For metastatic lung cancer, LRC is the local control of metastatic lung tumor here. Other patient demographic and clinical data, including age, gender; stage of disease, apatinib administered inclusion and withdrawal date, adverse events, oncologic clinical response, comorbid conditions, and smoking history, were retrieved from the CRIS database.

ELIGIBILITY:
Inclusion Criteria:

1. Between February 1, 2015 and May 19, 2018, 433 adult patients with gastric adenocarcinoma, lung adenocarcinoma and lung squamous cell carcinoma
2. Multiline chemotherapy failure and lack of standard treatment, received oral apatinib 250 mg daily at the Affiliated Hospital of Qingdao University.
3. Histologically proven were identified retrospectively using the Clinical Research Information Systems (CRIS) database.
4. All patients were with Karnofsky performance status over 70% or an Eastern Cooperative Oncology Group performance status of 0 to 1, with stable hepatic, hematologic, and renal functions.

Exclusion Criteria:

1. Cardiac disease and hemorrhagic disease were excluded.
2. Patients with lung cavitation before apatinib treated.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Between February 1, 2015 and May 19, 2018, 433 adult patients with gastric adenocarcinoma, lung adenocarcinoma and lung squamous cell carcinoma
  2. Multiline chemotherapy failure and lack of standard treatment, received oral apatinib 250 mg daily at the Affiliated Hospital of Qingdao University.
  3. Histologically proven were identified retrospectively using the Clinical Research Information Systems (CRIS) database.
  4. All patients were with Karnofsky performance status over 70% or an Eastern Cooperative Oncology Group performance status of 0 to 1, with stable hepatic, hematologic, and renal functions.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2018-05-19 (Actual); Study Completion 2018-05-19 (Actual)

PRIMARY OUTCOMES:
PFS (progression-free survival) | From February 1, 2015 to May 19, 2018 ,about 27 months
  Evaluation of the oncologic clinical response was based on the alternate, modified method. We concluded that incorporating an assessment of cavitation when measuring target lesions might more accurately reflect changes in tumor volume. It was used for target lesions in which the longest diameter of any cavitation (zero if no cavity presented) was subtracted from the longest total diameter of the lesion, with each measurement taken in the same plane, to provide an alternate measure that was used to calculate the sum of measurements for all target lesions.

SECONDARY OUTCOMES:
LRC (duration of locoregional control ) | From February 1, 2015 to May 19, 2018 , about 27 months
  For metastatic lung cancer, LRC is the local control of metastatic lung tumor here.